CLINICAL TRIAL: NCT03491436
Title: Pregnancy Remote Monitoring of Women at Risk for Gestational Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patient enrolled
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Wilfried Gyselaers, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRM-001
Record Dates: First submitted 2017-08-08; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Diabetic
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Women (at risk of) GDM will be included in this study. They receive a iHealth Align (a glucose monitor) and associated glycemiestrips.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote monitoring group (Experimental): Women (at risk of) GDM will be included in this study. They receive a iHealth Align (a glucose monitor) and associated glycemiestrips. The app of iHealth will be downloaded on the pregnant women's Smartphone to collect the data and to send them to the researcher in the hospital.
  Interventions: Device: iHealth Align

INTERVENTIONS:
Device: iHealth Align — remote monitor glucometer

SUMMARY:
Background: Remote monitoring (RM) is a new screenings- and or diagnostic tool in healthcare. In 2015, the PREMOM study (Pregnancy Remote Monitoring), in which patients with gestational hypertensive diseases did received a RM prenatal follow up, has started. The first results showed an added value of RM in the prenatal follow-up. Due to these results, a RM program for pregnant women with gestational diabetes mellitus (GDM) will be developed and evaluated.

Protocol: Women (at risk of) GDM will be included in this study. They receive a iHealth Align (a glucose monitor) and associated glycemiestrips. The app of iHealth will be downloaded on the pregnant women's Smartphone to collect the data and to send them to the researcher in the hospital.

The women is asked to perform four glycemie controls/day (sober and two hours after every mail) with the received glucose monitor. The monitor is connected via Wi-Fi and Bluetooth with the computer of the researches who controls and evaluated these data. Additionally, the pregnant women has to check daily her body weight with a weight scale of her own. They have to upload these data manually in the app on her smartphone.

When the pregnant women has an prenatal consultation, an overview with the data will be send to the responsible gynecologist. The gynecologist will also be alarmed when the pregnant women has three abnormal values at the same moment of the day (ex. Every morning after breakfast). When necessary, advice among life-style can be given or a referral to an endocrinologist can be made. The researches will not perform interventions by herself, only the responsible doctor can do this.

By analyzing the patients parameters when she's at home, a better vision can be achieved of the health of the mother and the child. This study will be conducted as a first research to get a better insight in the added value of RM in pregnancies complicated with GDM.

ELIGIBILITY:
Inclusion Criteria:

* women with confirmed GDM or at risk for this disease. Pregnancies > 10 weeks of gestation, primipara and multipara.

Exclusion Criteria:

* pregnancies < 10 weeks of gestation, congenital malformations of the fetus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose sober | an average of 30 weeks
  The women is asked to perform four glycemie controls/day (sober and two hours after every mail) with the received glucose monitor. The monitor is connected via Wi-Fi and Bluetooth with the computer of the researches who controls and evaluated these data.
  Has both mother and child advantages when the mother is screened and provided with the remote monitoring devices? is RM acceptable to use in the prenatal care for GDM and does it have in added value in gestational outcomes?
Weight once a day | an average of 30 weeks
  the pregnant women has to check daily her body weight with a weight scale of her own. They have to upload these data manually in the app on her smartphone.
  Has both mother and child advantages when the mother is screened and provided with the remote monitoring devices? is RM acceptable to use in the prenatal care for GDM and does it have in added value in gestational outcomes?
blood glucose 2 hours after meal 1 | an average of 30 weeks
  The women is asked to perform four glycemie controls/day (sober and two hours after every mail) with the received glucose monitor. The monitor is connected via Wi-Fi and Bluetooth with the computer of the researches who controls and evaluated these data.
  Has both mother and child advantages when the mother is screened and provided with the remote monitoring devices? is RM acceptable to use in the prenatal care for GDM and does it have in added value in gestational outcomes?
blood glucose 2 hours after meal 2 | through study completion
  The women is asked to perform four glycemie controls/day (sober and two hours after every mail) with the received glucose monitor. The monitor is connected via Wi-Fi and Bluetooth with the computer of the researches who controls and evaluated these data.
  Has both mother and child advantages when the mother is screened and provided with the remote monitoring devices? is RM acceptable to use in the prenatal care for GDM and does it have in added value in gestational outcomes?
blood glucose 2 hours after meal 3 | an average of 30 weeks
  The women is asked to perform four glycemie controls/day (sober and two hours after every mail) with the received glucose monitor. The monitor is connected via Wi-Fi and Bluetooth with the computer of the researches who controls and evaluated these data.
  Has both mother and child advantages when the mother is screened and provided with the remote monitoring devices? is RM acceptable to use in the prenatal care for GDM and does it have in added value in gestational outcomes?

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided